CLINICAL TRIAL: NCT04965597
Title: Hematopoietic Cell Transplantation Using Treosulfan-Based Conditioning for the Treatment of Bone Marrow Failure Diseases
Brief Title: Treosulfan-Based Conditioning Regimen Before a Blood or Bone Marrow Transplant for the Treatment of Bone Marrow Failure Diseases (BMT CTN 1904)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1904; 2U10HL069294-11 (NIH); RG1121820 (Other: Fred Hutch/University of Washington Cancer Consortium); 10840 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-13862 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-21; First posted 2021-07-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Bone Marrow Failure Syndrome; Congenital Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Hereditary Sideroblastic Anemia; Paroxysmal Nocturnal Hemoglobinuria; Shwachman-Diamond Syndrome; Hematologic Neoplasm With Germline GATA2 Mutation; Hematologic Neoplasm With Germline SAMD9 Mutation; Hematologic Neoplasm With Germline SAMD9L Mutation
Keywords: Bone Marrow Failure Disorders; HSCT; Treosulfan; Unrelated donor; Matched donor; mismatched donor; transplant
MeSH Terms: conditions — Bone Marrow Failure Disorders; Congenital amegakaryocytic thrombocytopenia; Anemia, Diamond-Blackfan; Anemia, Hypochromic; Hemoglobinuria, Paroxysmal; Shwachman-Diamond Syndrome | interventions — treosulfan; fludarabine phosphate; Tacrolimus; Methotrexate; Antilymphocyte Serum; thymoglobulin; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (conditioning regimen; transplant; GVHD prophylaxis) (Experimental): CONDITIONING REGIMEN: Patients receive treosulfan IV over 120 minutes on days -6 to -4, fludarabine phosphate IV over 60 minutes on days -6 to -2, and rATG IV over 4-6 hours on days -4 to -2.
  TRANSPLANTATION: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously beginning on day -2 and a taper beginning on day 180. Patients may also receive tacrolimus PO. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Patients undergo ECHO or MUGA as well as possible x-ray or CT at baseline and undergo bone marrow biopsy and aspiration at baseline and follow up. Patients also undergo blood sample collection throughout the trial.
  Interventions: Drug: Treosulfan; Drug: Fludarabine Phosphate; Drug: Tacrolimus; Drug: Methotrexate; Biological: Lapine T-Lymphocyte Immune Globulin; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Bone Marrow Transplantation; Other: Quality-of-Life Assessment; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection; Procedure: X-Ray Imaging; Procedure: Computed Tomography

INTERVENTIONS:
Drug: Treosulfan — Given IV
  Other Names: Dihydroxybusulfan; Ovastat; Treosulphan; Tresulfon; Trecondi
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; 9H-purin-6-amine; 2-fluoro-9-(5-O-phosphono-beta-D-arabinofuranosyl); Beneflur; Fludara; Fludarabine-5'-Monophosphate; SH T 586
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; Emthexat; Emtexate; Farmitrexat; Methotrexate LPF; Methylaminopterin; Methotrexatum; Metotrexato; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-Thymocyte Globulin Rabbit; Grafalon; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; rATG; Thymoglobulin; Antithymocyte globulin rabbit ATG; Imtix
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Procedure: Allogeneic Bone Marrow Transplantation — Undergo bone marrow transplant
  Other Names: Allo BMT; Allogeneic Blood and Marrow Transplantation; Allogeneic BMT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; Multi-Gated Acquisition Scan; MUGA Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology
Procedure: Computed Tomography — Undergo chest CT
  Other Names: Computed Axial Tomography; CAT Scan; CT Scan

SUMMARY:
This phase II trial tests whether treosulfan, fludarabine, and rabbit antithymocyte globulin (rATG) work when given before a blood or bone marrow transplant (conditioning regimen) to cause fewer complications for patients with bone marrow failure diseases. Chemotherapy drugs, such as treosulfan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Fludarabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. rATG is used to decrease the body's immune response and may improve bone marrow function and increase blood cell counts. Adding treosulfan to a conditioning regimen with fludarabine and rATG may result in patients having less severe complications after a blood or bone marrow transplant.

DETAILED DESCRIPTION:
OUTLINE:

CONDITIONING REGIMEN: Patients receive treosulfan intravenously (IV) over 120 minutes on days -6 to -4, fludarabine phosphate IV over 60 minutes on days -6 to -2, and lapine T-lymphocyte immune globulin (rATG) IV over 4-6 hours on days -4 to -2.

TRANSPLANTATION: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously beginning on day -2 and a taper beginning on day 180. Patients may also receive tacrolimus orally (PO). Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) as well as possible chest radiography (x-ray) or computed tomography (CT) at baseline and undergo bone marrow biopsy and aspiration at baseline and follow up. Patients also undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 1 year from transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 1.0 year of age and less than 50.0 years of age at the time of enrollment (i.e. patient must have celebrated their 1st birthday when enrolled and must NOT have celebrated their 50th birthday when enrolled; 49.99 years)
* Underlying BMFD treatable by allogenic HCT
* Shwachman-Diamond syndrome

  * Criteria for Diagnosis:

    * A pathogenic mutation(s) for Shwachman-Diamond syndrome
    * For those patients tested but lacking a genetic mutation they must meet both *** criteria below:

      * Exocrine pancreatic dysfunction as defined by at least one of the following:

        * Pancreatic isoamylase below normal (age >= 3 years old), OR
        * Fecal elastase < 200, AND
      * Bone marrow failure as evidence by at least one of the following:

        * Intermittent or persistent neutropenia (absolute neutrophil count < 1,500/uL), OR
        * Hypo-productive anemia with a hemoglobin concentration below the age-related adjusted norms, OR
        * Unexplained macrocytosis, OR
        * Platelet count < 150,000/uL without alternative etiology, OR
        * Hypocellular bone marrow
  * Indications for HCT:

    * Severe neutropenia (absolute neutrophil count [ANC] < 500/uL), OR
    * Severe anemia (hemoglobin < 8 g/dL) or transfusion-dependent anemia, OR
    * Severe thrombocytopenia (platelet count < 20,000/uL) or transfusion-dependent thrombocytopenia, OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 eligibility review committee (ERC). In addition, patients with severe or recurrent infections will be reviewed by the ERC if they do not meet the indications for transplant listed above
* Diamond Blackfan Anemia

  * Criteria for Diagnosis:

    * A pathogenic mutation for Diamond Blackfan anemia
    * For those patients tested but lacking a genetic mutation the patient must meet the first *** criteria and at least one of the subsequent *** criteria listed below:

      * History of deficiency of erythroid precursors in an otherwise cellular bone marrow AND,
      * Reticulocytopenia, OR
      * Elevated adenosine deaminase activity, OR
      * Elevated hemoglobin F, OR
      * Macrocytosis, OR
      * Congenital anomalies
  * Indications for HCT:

    * Red blood cell (RBC) transfusion dependent anemia despite an adequate trial of steroids; OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC
* Congenital Sideroblastic anemia

  * Criteria for Diagnosis:

    * A pathogenic mutation(s) for sideroblastic anemia
    * For those patients tested but lacking a genetic mutation:

      * Presence of ringed sideroblasts in the bone marrow excluding acquired causes of ringed sideroblasts such as lead poisoning & zinc toxicity
  * Indications for HCT:

    * Severe anemia (hemoglobin < 8 g/dL) or transfusion-dependent anemia OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC
* GATA2 mutation with associated marrow failure

  * Criteria for Diagnosis:

    ** A pathogenic mutation(s) for GATA2
  * Indications for HCT:

    * Severe neutropenia (ANC < 500/uL), OR
    * Severe anemia (hemoglobin < 8 g/dL) or transfusion-dependent anemia, OR
    * Severe thrombocytopenia (platelet count < 20,000/uL) or transfusion-dependent thrombocytopenia, OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC. In addition, patients with severe or recurrent infections will be reviewed by the ERC if they do not meet indications for transplant listed above
* SAMD9 or SAMD9L disorders

  * Criteria for Diagnosis:

    ** A pathogenic mutation(s) for SAMD9 or SAMD9L
  * Indications for HCT:

    * Severe neutropenia (ANC < 500/uL), OR
    * Severe anemia (hemoglobin < 8 g/dL) or transfusion-dependent anemia, OR
    * Severe thrombocytopenia (platelet count < 20,000/uL) or transfusion-dependent thrombocytopenia, OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC
* Congenital amegakaryocytic thrombocytopenia

  * Criteria for Diagnosis:

    * A pathogenic mutation(s) for congenital amegakaryocytic thrombocytopenia.
    * For those patients tested but lacking a genetic mutation the patient must meet criteria below:

      * Thrombocytopenia early in life, AND
      * History of bone marrow demonstrating megakaryocyte hypoplasia
  * Indications for HCT:

    * Severe thrombocytopenia (platelet count < 20,000/uL) or transfusion-dependent thrombocytopenia, OR
    * Neutropenia defined as an ANC < 500/uL, OR
    * Severe anemia (hemoglobin < 8 g/dL) or transfusion-dependent anemia, OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC
* Paroxysmal nocturnal hemoglobinuria

  * Criteria for Diagnosis:

    * Paroxysmal nocturnal hemoglobinuria (PNH) clone size in granulocytes >= 10%, AND
    * Complement mediated intravascular hemolysis with an elevated LDH (above institutional upper limits of normal)
  * Indications for HCT:

    * PNH with thrombosis despite adequate medical management, OR
    * PNH with intravascular hemolysis requiring transfusion support despite adequate medical management, OR
    * Additional clinical or laboratory data may be considered for protocol eligibility following review by protocol 1904 ERC. In addition, patients with PNH and cytopenias may be considered for the protocol eligibility following review by protocol 1904 ERC
* An undefined BMFD: a patient with a BMFD for whom a genetic mutation responsible for their bone marrow failure phenotype has not been identified (excluding PNH) will be eligible for this clinical trial following approval by Blood and Marrow Transplant Clinical Trials Network (BMT CTN) 1904 ERC

  * A BMFD with a known genetic mutation but not listed above will be eligible for this clinical trial following approval by BMT CTN 1904 ERC
* Patient and/or legal guardian must sign informed consent prior to initiation of conditioning for BMT CTN 1904
* Note: The following patients MUST be reviewed by the BMT CTN 1904 ERC in order to determine if they are eligible for this trial:

  * All patients with Shwachman-Diamond syndrome, Diamond Blackfan anemia, congenital sideroblastic anemia, and congenital amegakaryocytic thrombocytopenia who have had genetic testing and a genetic mutation responsible for their disease was not identified
  * All patients with an undefined BMFD: a patient with a BMFD for whom a genetic mutation responsible for their bone marrow failure phenotype has not been identified, excluding PNH
  * All patients with a BMFD and a known genetic mutation that is not listed above
  * All patients with GATA2 mutation and associated marrow failure
  * All patients with SAMD9 or SAMD9L disorders
  * There may be circumstances where a treating physician will consider a transplant for a patient with a BMFD who does not meet all the criteria listed under "indications for HCT". In these situations, treating physicians may submit their patient to the BMT CTN 1904 ERC for review in order to determine if the patient is eligible for this clinical trial based on additional clinical or laboratory information
  * Many patients with BMFD can have bone marrow evaluations that raise concern for possible myelodysplastic syndrome (MDS) including but not limited to dysplastic bone marrow evaluations or cytogenetic abnormalities. However, in patients BMFD these findings are not necessarily diagnostic or consistent with MDS. Therefore, given the complexities of diagnosing MDS in patients with BMFD, all patients with bone marrow evaluations concerning for possible MDS should be submitted to the ERC for review to confirm or exclude MDS. This is particularly important as we do not want to exclude potentially eligible patients due to an incorrect diagnosis of MDS
* HLA-MATCHED RELATED DONOR: HLA-matched sibling: Must be a minimum HLA-6/6 matched to the recipient at HLA-A, -B (serologic typing) and DRB1 (high-resolution typing)
* HLA-MATCHED RELATED DONOR: HLA-matched related (phenotypic match): Fully matched for HLA-A, -B, -C, -DRB1, and DQB1 by high-resolution typing.
* HLA-MATCHED RELATED DONOR: If a genetic mutation is known for the patient, the HLA-matched related donor [either HLA-matched sibling or HLA-matched related (phenotypic match)] must be screened for the same genetic mutation if clinically appropriate and should be confirmed to not have the same genetic disease (this does not include patients with PNH). Consult the protocol team with questions
* HLA-MATCHED RELATED DONOR: If a patient has an undefined BMFD (a patient with a BMFD for whom a genetic mutation responsible for their bone marrow failure phenotype has not been identified), the HLA-matched related donor [either HLA-matched sibling or HLA-matched related (phenotypic match)] must have an evaluation as directed by the treating physician to confirm that the donor does not have the same underlying disease. This will include a complete blood count (CBC) with differential and potentially a bone marrow evaluation or other studies as directed by the treating physician
* UNRELATED DONOR: Fully matched for HLA-A, -B, -C, -DRB1, and DQB1 by high-resolution typing OR
* UNRELATED DONOR: Mismatched for a single HLA-class 1 allele (HLA-A, -B, or -C) by high-resolution typing; OR
* UNRELATED DONOR: Mismatched for a single HLA DQB1 allele or antigen by high-resolution typing

  * Note: donor patient (DP) matching per institutional practice
* DONOR SELECTION RECCOMENDATIONS: in the case where there are multiple donor options, donors should be selected based on the following priority numbered below:

  * Unaffected fully HLA-matched sibling
  * Unaffected fully phenotypically HLA-matched related donor
  * Fully HLA-matched unrelated donor
  * Unrelated donor with single allele or antigen level mismatch at DQB1
  * Unrelated donor with single allele level mismatch at class 1 (HLA-A, -B, or -C)

Exclusion Criteria:

* Patients with idiopathic aplastic anemia, Fanconi anemia, dyskeratosis congenita, and congenital neutropenia
* Patients with MDS as defined by the World Health Organization (WHO) or leukemia
* Prior allogeneic HCT
* Patient's weight =< 10.0 kg (actual body weight and adjusted body weight) at time of study enrollment
* Lansky (patients < 16 years of age) or Karnofsky (patients >= 16 years of age) performance < 70%
* Left ventricular ejection fraction < 50% by echocardiogram or multi-gated acquisition (MUGA) scan

  * For patients unable to obtain a left ventricular ejection fraction, left ventricular shortening fraction of < 26%
* Diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected/adjusted for hemoglobin) < 50%, forced expiratory volume (FEV)1 < 50% predicted, and forced vital capacity (FVC) < 50% predicted
* For patients unable to perform pulmonary function tests (PFTs) due to age or developmental delay: oxygen (O2) saturation < 92% on room air
* On supplemental oxygen
* Estimated creatinine clearance < 60 mL/minute/1.73m^2 (estimated per institutional practice)
* Dialysis dependent
* Conjugated bilirubin > 2 x upper limit of normal for age (ULN, unless attributable to Gilbert's syndrome)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 4 x ULN for age, or
* Fulminant liver failure or cirrhosis
* Iron overload - This exclusion criterion only applies to patients who are considered at risk for hepatic or cardiac iron overload. Therefore, not all patients enrolled on this protocol will undergo formal hepatic or cardiac iron assessment

  * For patients with a history of significant transfusions defined as >= 8 packed red blood cell transfusions per year for >= 1 year or have received >= 20 packed red blood cell transfusions (lifetime cumulative) will require formal hepatic and cardiac iron measurement. In addition, patients with a prior history of hepatic or cardiac iron overload will also require formal assessment for iron overload. Patients are excluded if:
  * Hepatic iron content >= 8 mg Fe/g dry weight by liver magnetic resonance imaging (MRI) using a validated methodology (such as T2 * MRI or ferriscan) or liver biopsy per institutional practice
  * Cardiac iron content < 25 msec by cardiac T2 * MRI
* Uncontrolled bacterial infection within 1 week of study enrollment. Uncontrolled is defined as currently taking medication with no clinical improvement or progression on adequate medical treatment
* Uncontrolled viral or fungal infection within 30 days of study enrollment. Uncontrolled is defined as currently taking medication with no clinical improvement or progression on adequate medical treatment
* Positive for human immunodeficiency virus (HIV)
* Presence of clinically significant anti-donor human leukocyte antigen (HLA)-antibodies per institutional practice
* Prior solid organ transplant
* Patients with prior malignancies except resected non-melanoma skin cancer or treated cervical carcinoma in situ
* Females who are pregnant or breast-feeding
* Females and males of childbearing potential who are unwilling to practice an effective method of contraception or agree to abstinence from the time of signing informed consent through 12 months post-transplant or off tacrolimus whichever is later
* Known hypersensitivity to treosulfan or fludarabine
* Known life-threatening reaction (i.e. anaphylaxis) to Thymoglobulin that would prohibit use for the patient as this study requires use of the Thymoglobulin preparation of anti-thymocyte globulin (ATG)

Ages: 1 Year to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Graft-Versus Host-Disease (GVHD)-Free Event-Free Survival (EFS) | 1 year post-HCT
  The primary endpoint is the incidence of 1-year GVHD free, EFS (GEFS). An event is defined as death due to any cause, primary or secondary graft failure/rejection, or 2nd HCT whichever occurs first. Grade III-IV acute GVHD and chronic GVHD (using National Institutes of Health [NIH] consensus criteria) requiring systemic immune suppression will be considered in this estimate.

SECONDARY OUTCOMES:
Overall Survival | Day 100 post-HCT
  Overall survival at day 100 after HCT
Overall Survival | 6 months post-HCT
  Overall survival at 6 months after HCT
Overall Survival | 1 year post-HCT
  Overall survival at 1 year after HCT
Event-Free Survival | 1 year post-HCT
  Event-free survival will be estimated at 12 months after HCT. An event is defined as death due to any cause, primary or secondary graft failure/rejection, or 2nd HCT, whichever occurs first
Hematologic Recovery: Neutrophil recovery | Assessed up to 1 year post-HCT
  Hematologic recovery will be assessed according to neutrophil recovery after transplant. Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) ≥ to 500/mm3 for 3 consecutive measurements on 3 different days. The first of the three days will be designated the day of neutrophil recovery. The competing event is death without neutrophil recovery.
Hematologic Recovery: Platelet recovery | Day 100 post-HCT
  Hematologic recovery will be assessed according to platelet counts recovery after transplant. Platelet recovery is defined as the first day of a minimum of 3 days that the patient has a sustained platelet count ≥ 20,000/mm3 with no platelet transfusions in the preceding 7 days. The first day of sustained platelet count above these thresholds will be designated the day of platelet engraftment.
Donor Chimerism (CD3 and Myeloid) | Day 28 post-HCT
  Proportions of patients with full (>95%), mixed (5-95%), or rejection (<5%) myeloid
Donor Chimerism (CD3 and Myeloid) | Day 100 post-HCT
  Proportions of patients with full (>95%), mixed (5-95%), or rejection (<5%) myeloid
Donor Chimerism (CD3 and Myeloid) | 1 year post-HCT
  Proportions of patients with full (>95%), mixed (5-95%), or rejection (<5%) myeloid
Primary graft failure/rejection | Day 42 post-HCT
  Defined as never achieving ANC ≥ 500/μL or never achieving ≥ 5% donor myeloid chimerism assessed by peripheral blood chimerism assays by day +42 post-HCT. Second infusion of hematopoietic cells is also considered indicative of primary graft failure by day +42 post-HCT
Secondary graft failure/rejection post-HCT | Assessed up to 1 year post-HCT
  Defined as < 5% donor myeloid chimerism in peripheral blood beyond day +42 post-HCT in patients with prior documentation of hematopoietic recovery with ≥ 5% donor cells by day +42 post-HCT. Second infusion of hematopoietic cells is also considered indicative of secondary graft failure.
Grade II-IV and grade III-IV GVHD at day 100 | Day 100 post-HCT
  The cumulative incidences of acute grade II-IV and III-IV GVHD at day 100 after HCT will be determined.
Grade II-IV and grade III-IV GVHD at day 180 | Day 180 post-HCT
  The cumulative incidences of acute grade II-IV and III-IV GVHD at day 100 after HCT will be determined.
Chronic GVHD | 1 year post-HCT
  The cumulative incidence of chronic GVHD (using NIH consensus criteria) requiring systemic immune suppression at 1 year after HCT will be determined. Data will be collected directly from providers and chart review as defined by the NIH Consensus Conference Criteria
Incidence of grade 3-5 toxicities | Day 30 post-HCT
  Grade 3-5 toxicities by day 30 after HCT
Incidence of grade 3-5 toxicities | Day 100 post-HCT
  Grade 3-5 toxicities by day 100 after HCT
Incidence of grade 2-3 systemic infections | 6 months post-HCT
  All microbiologically documented infections or significant infections requiring antibiotic/antifungal therapy occurring up to 6 months after HCT
Incidence of Epstein Barr virus (EBV) reactivation requiring therapy | Day 180 post-HCT
  The incidence of EBV reactivation requiring therapy in the first 180 days after HCT, and of EBV-associated lymphoproliferative disorder in the first 180 days after HCT will be evaluated.
Incidence of EBV-associated lymphoproliferative disorder | Day 180 post-HCT
Incidence of cytomegalovirus (CMV) reactivation requiring therapy by day 180 post-HCT | Up to day 180 post-HCT

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Burroughs, MD, Study Chair — Fred Hutch/University of Washington Cancer Consortium; Margaret MacMillan, MD, Study Chair — University of Minnesota
Locations (24):
- United States (24):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital/UCSD, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cohen Children's Hospital of NY, Queens, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's/University of Utah, Salt Lake City, Utah
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT04965597/ICF_000.pdf